CLINICAL TRIAL: NCT01430702
Title: Feasibility of Using a Telemedicine Medication Delivery Unit for Older Adults That Require Medication Assistance During Transition Form Hospital to Home
Brief Title: Feasibility of Using a Telemedicine Medication Delivery Unit for Older Adults
Acronym: EMMA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FY2010-007
Record Dates: First submitted 2011-09-01; First posted 2011-09-08 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Medication Adherence; Medication Nonadherence; Adverse Reaction to Drug
MeSH Terms: conditions — Medication Adherence; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computerized medication delivery unit (Experimental): Those hospitalized patients that meet all inclusion and exclusion criteria will be provided with a computerized medication delivery unit for use in their homes for the 30-day period following discharge.
  Interventions: Device: Computerized medication delivery unit (Electronic Medication Management Assistant (EMMA)

INTERVENTIONS:
Device: Computerized medication delivery unit (Electronic Medication Management Assistant (EMMA) — The patient's prescriptions and refills are packaged in standard-sized blister cards and loaded into EMMA units. The EMMMA identifies each medication automatically - no patient input is required. When activated by the patient, the medications are selected from the blister cards and released into the delivery tray. The EMMA will remain in the patient's home for a period of 30-days immediately following hospitalization. After 30 days, the EMMA MDU will become available for the next eligible patient. This maximizes the number of patients that can benefit from the MDU, while addressing the transition period when medication-reconciliation problems are most common.
  Other Names: Electronic Medication Management Assistant (EMMA)

SUMMARY:
Care transition interventions have been successful in reducing medication-related problems and associated rehospitalization primarily by focusing on medication reconciliation conducted by trained healthcare professionals. Programs to improve the medication reconciliation process have largely been effective, but have limitations including the expense associated with recruiting, training, and retaining care transition healthcare professionals (e.g., nurses and nurse practitioners) the ability to provide services within a finite geographic area, and the retrospective nature of the reconciliation process which usually occurs in the home following hospital discharge. Our short-term objective is to use Pennsylvania Department of Aging resources to assess the feasibility of using a telemedicine medication delivery unit for frail older adults that require medication assistance in their home immediately following an acute hospitalization. As part of this feasibility assessment, the investigators will assess (1) recruitment process and procedures, (2) data collection procedures, (3) resource utilization, (4) drop-out rates, (5) acceptability and usability of the EMMA® telemedicine medication delivery unit, (6) medication adherence, and (7) medication-reconciliation errors during transition from hospital to home.

DETAILED DESCRIPTION:
Care transition interventions have been successful in reducing medication-related problems and associated re-hospitalization primarily by focusing on medication reconciliation conducted by trained healthcare professionals. Medication reconciliation is the process of identifying discrepancies in drug regimens prescribed in different care settings or at different time points within the same setting, to inform prescribing decisions and prevent medication-related problems, including medication errors (MEs) and adverse drug events (ADEs). MEs and ADEs are particularly common during and following hospitalization, when multiple changes to a patients' medication regimens may be accompanied by inadequate patient education,\ follow-up, and continuity of care with primary care physicians and case managers. As a result of these problems, as many as 42% of general medical patients experience an ME or ADE after hospital discharge, with disproportionate impacts on older adults with chronic medical conditions. Post-hospital ADEs can be expensive, as12% result in an emergency department evaluation and 5% in readmission, which is associated with a significant increase in healthcare resource utilization and further fragmentation in care.

Programs to improve the medication reconciliation process have largely been effective, but have limitations including the expense associated with recruiting, training, and retaining care transition healthcare professionals (e.g., nurses and nurse practitioners), the ability to provide services within a finite geographic area, and the retrospective nature of the reconciliation process, which usually occurs in the home following hospital discharge. The investigators short-term objective is to use Pennsylvania Department of Aging resources to assess the feasibility of using a telemedicine medication delivery unit for frail older adults that require medication assistance in their home immediately following an acute hospitalization. As part of this feasibility assessment, the investigators will assess several methods and intervention-related components.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 65 years of age.
* Admitted during the study period for a nonpsychiatric condition to UPMC Presbyterian Hospital.
* Documented in their medical record at least 1 of 11 diagnoses, including: stroke, congestive heart failure, coronary artery disease, cardiac arrhythmias, chronic obstructive pulmonary disease, diabetes mellitus, spinal stenosis, hip fracture, peripheral vascular disease, deep venous thrombosis, and pulmonary embolism.
* Prescribed > 5 and < 20 regularly scheduled (i.e., non-PRN) prescription medications.
* Be from and return to a home setting (not assisted living, skilled nursing, program for all-inclusive care of the elderly, etc).
* Reside within a predefined geographic radius (i.e., Allegheny, Beaver, Butler, Fayette, Washington or Westmoreland Counties) of the hospital.
* Have a working telephone.
* Be English speaking.
* Have an informal caregiver or support person.

Exclusion Criteria:

* Have an active prescription for narcotic analgesic.
* Enrolled in or plan to enroll into hospice.
* Plans to travel in the next 30 days.
* Participating in another research protocol.
* Have evidence in the chart of a diagnosis of active delirium.
* Have evidence in the chart of a diagnosis of dementia.
* Have evidence in the chart of legal blindness.
* Unable to demonstrate appropriate use of the EMMA medication delivery unit.
* Unable to receive ATT wireless services data plan based on physical address.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
medication adherence | 30-day
  The investigators will assess adherence by determining the number of regularly scheduled medications taken vs. prescribed (data will come from the EMMA® Report software).

SECONDARY OUTCOMES:
medication-reconciliation errors during transition from hospital to home | 30-day
  Finally, the investigators will measure medication-reconciliation errors using the Medication Discrepancy Tool (MDT).
acceptability and usability of the EMMA® telemedicine medication delivery unit | 30-day
  The investigators will assess acceptability and usability of the EMMA® telemedicine medication delivery unit through a previously validated instrument developed by the The Quality of Life Technology (QoLT) Center at Carnegie Mellon University.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Handler, MD, PhD, CMD, Principal Investigator — University of Pittsburgh -- of the Commonwealth System of Higher Education
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States